CLINICAL TRIAL: NCT00481845
Title: Randomized Phase 2 Trial of Anastrozole Combined With Novel Agent ZD6474 in the Neoadjuvant Treatment of Postmenopausal Patients With Hormone Receptor-Positive Breast Cancer
Brief Title: Phase 2 Anastrozole and Vandetanib (ZD6474) in Neoadjuvant Treatment of Postmenopausal Hormone Receptor-Positive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Stanford University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Mark Pegram, Susy Yuan-Huey Hung Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-08051; BRSADJ0008 (Other: OnCore); 97923 (Other: Stanford University Alternate IRB Approval Number)
Record Dates: First submitted 2007-05-31; First posted 2007-06-04 (Estimated); Results first posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — vandetanib; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vandetanib + Anastrozole (Experimental): Vandetanib and Anastrozole as neoadjuvant therapy
  Interventions: Drug: Vandetanib; Drug: Anastrozole
- Anastrozole (Active Comparator): Anastrozole as neoadjuvant therapy
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Vandetanib — 300 mg daily
  Other Names: Zactima; ZD6474
  Arms: Vandetanib + Anastrozole
Drug: Anastrozole — 1 mg daily
  Other Names: Arimidex

SUMMARY:
In this study we plan to study the combination of ZD6474, a dual inhibitor of EGFR and VEGFR-2 with anastrozole in the neoadjuvant setting for patients with Stage I-III breast cancer. The aim is to overcome mechanisms of resistance and simultaneously block multiple critical signaling pathways known to stimulate breast cancer.

DETAILED DESCRIPTION:
The use of adjuvant chemotherapy and endocrine therapy has had a significant impact on breast cancer survival. However, not all patients will benefit from each of these therapies. Increasing data suggests that patients with hormone receptor-positive breast cancer derive marginal benefit from the addition of adjuvant chemotherapy. Identification and characterization of cellular signaling pathways active in the pathogenesis of breast cancer has lead to the development of multiple targeted therapies that hold enormous promise for patients with less toxicity than conventional chemotherapy. Treatment strategies employing neoadjuvant therapy have found that pCR is predictive for ultimate outcome. Due to this, the use of neoadjuvant therapy has become an intense area of investigation in operable breast cancer. In the IMPACT trial, the aromatase inhibitor anastrozole was found to improve eligibility for breast conservation and was associated with a favorable clinical objective response after 12 weeks of therapy.

In this proposed study, we plan to study the combination of ZD6474, a dual inhibitor of EGFR and VEGFR-2, with anastrozole in the neoadjuvant setting for patients with Stage I-III breast cancer. The aim is to overcome mechanisms of resistance and simultaneously block multiple critical signaling pathways known to stimulate breast cancer. The two agents have non-overlapping toxicities and are both administered orally, allowing for a more tolerable treatment regimen. By using this combination in the neoadjuvant setting, we will target the critical signaling pathways early and follow tumor responses during therapy, allowing for prompt evaluation of the effectiveness of this treatment strategy. Pathologic tumor specimens obtained at the time of definitive surgery will be evaluated for pathologic complete response thus adding to the body of literature. By examining molecular markers such as ER, PR, EGFR, and Ki-67 pre- and post-treatment, we hope to correlate modulations in these biomarkers to response. Finally, using a novel second generation functional breast MRI we will investigate the ability of MRI to predict response to antiangiogenic therapy.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed invasive, hormone receptor-positive (ER and/or PR positive) breast cancer

* Stage I-III breast cancer including any primary tumor ≥ 1 cm by ultrasound
* Diagnosis by core needle biopsy with placement of metallic clip at tumor site
* Sentinel lymph node biopsy (US-guided FNA may be substituted if palpable axillary lymphadenopathy)
* Evaluation by a surgeon to determine eligibility for breast conservation
* Postmenopausal status (age ≥ 60 yo; or < 60 yo and FSH and estradiol in the postmenopausal range, prior bilateral oophorectomy)
* Serum creatinine < 1.5 x upper limit of normal (ULN) or creatinine clearance > 50 mL/minute (calculated by Cockcroft-Gault formula.)
* Serum bilirubin < 1.5 x ULN
* Serum potassium ≥ 4 mmol/L (supplementation allowed)
* Serum calcium or magnesium within normal range (supplementation allowed)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5 x ULN or alkaline phosphatase (ALP) ≤ 2.5 x ULN
* ECOG Performance Status 0,1,2
* ECG QTc < 480 msec
* Measurable disease
* Written, informed consent

Exclusion Criteria:- Inflammatory breast cancer

* Metastatic breast cancer excluding disease in regional lymph nodes
* Inoperable disease considered irreversible with neoadjuvant endocrine therapy
* HER2-overexpressed breast cancer
* Prior chemotherapy or radiotherapy for the treatment of the current breast cancer
* Prior hormonal therapy for the treatment of the current breast cancer
* Prior surgical biopsy, lumpectomy, mastectomy for the current breast cancer
* Any concurrent condition which in the Investigator's opinion makes it inappropriate for the patient to participate in the trial or which would jeopardize compliance with the protocol
* Currently active diarrhea that may affect the ability of the patient to absorb ZD6474 or tolerate diarrhea
* Clinically significant cardiac event such as myocardial infarction; New York Heart Association (NYHA) classification of heart disease >2 within 3 months before entry; or presence of cardiac disease that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia.
* History of arrhythmia (multifocal premature ventricular contractions (PVCs), bigeminy, trigeminy, ventricular tachycardia (VT) or uncontrolled atrial fibrillation) which is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained VT. Atrial fibrillation controlled on medication is not excluded.
* Previous history of QTc prolongation as a result of another medication that required discontinuation of that medication.
* Congenital long QT syndrome or 1st degree relative with unexplained sudden death < 40 years of age.
* Presence of left bundle branch block (LBBB).
* QTc with Bazett's correction that is unmeasurable, or ≥ 480 msec on screening ECG. If a patient has QTc ≥ 480 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be < 480 msec in order for the patient to be eligible for the study.
* Use of any concomitant medication that may cause QTc prolongation, induce Torsades de Pointes or induce CYP3A4 function.
* Hypertension not controlled by medical therapy (systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mm hg).
* Previous or current malignancies of other histologies within the last 5 years, with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin.
* Major surgery within 4 weeks or incompletely healed surgical incision before starting study therapy.
* Receipt of any investigational agents within 30 days prior to commencing study treatment
* Previous enrollment or randomization of treatment in the present study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Pegram, MD, Principal Investigator — Stanford Cancer Institute, Stanford University Medical Center
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vandetanib + Anastrozole | Anastrozole
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vandetanib + Anastrozole | Anastrozole | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Tumor Objective Response by MRI
Description: Determine tumor objective response rate by MRI. (CR): Disappearance of the target lesion (PR): At least a 30% decrease in the longest diameter of the target lesion taking as reference the baseline LD (PD): At least a 20% increase in the LD of target lesion, taking as reference the baseline LD or the appearance of one or more new lesions (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the baseline LD.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Vandetanib + Anastrozole | Anastrozole
Number analyzed (Participants) | 1 | 0
Participants
  Complete Response- CR | 0 | 0
  Partial Response- PR | 0 | 0
  Progressive Disease- PD | 0 | 0
  Stable Disease-SD | 1 | 0

2. Secondary Outcome: Pathologic Complete Response
Time Frame: 1 year
Population: CR+PR
Measure: Count of Participants; unit: Participants
Arm/Group | Vandetanib + Anastrozole | Anastrozole
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: All AEs or SAEs collected during the 4 months (12 cycles) span on treatment
Arm/Group | Vandetanib + Anastrozole | Anastrozole
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vandetanib + Anastrozole (N=1) | Anastrozole (N=0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hypertension (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vandetanib + Anastrozole (N=1) | Anastrozole (N=0)
Vague chest discomfort (Cardiac disorders) | 1 (2) | 0 (0)
Sweaty palms (Nervous system disorders) | 1 (1) | 0 (0)
Painic attack (Nervous system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
increasing reflux symptoms (Gastrointestinal disorders) | 1 (1) | 0 (0)
Onset asthma symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
esophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No